CLINICAL TRIAL: NCT00153153
Title: Extended Use of Polyethyleneglycol3350 Laxative in Constipated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 851-CR1
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

INTERVENTIONS:
Drug: polyethyleneglycol3350

SUMMARY:
To evaluate the safety and efficacy of extended use of polyethyleneglycol3350 laxative as compared to placebo in constipated patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age
* Constipated according to ROME I criteria
* On average, fewer than 3 satisfactory BMs per week during the observation period
* If female and of childbearing potential, patient must be surgically sterilized or using oral contraceptives, depot contraceptives, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so during the duration of study
* Are otherwise in good health, as judged by a physical examination
* In the investigator's judgment, patient is mentally competent to sign an instrument of informed consent

Exclusion Criteria:

* Patients with heme positive stool at screening. Patients with heme positive stool that can be attributed to hemorrhoids or anal fissures are eligible for inclusion.
* Patients with hypo- or hyperthyroidism as determined by history, or screening TSH results.
* Patients with known or suspected perforation or obstruction.
* History of gastric retention, inflammatory bowel disease, bowel resection, or colostomy.
* Patients with a known history of organic cause for their constipation.
* Patients meeting the ROME definition of Irritable Bowel Syndrome
* Patients currently taking any of the following medications that are known to effect bowel habits:

  * Antidiarrheals
  * Antacids containing magnesium or aluminum salts
  * Anticholinergics
  * Antispasmodic agents
  * Erythromycin and other macrolides
  * Octreotide
  * Lotronex, Zofran, or other 5-HT3 antagonists
  * Zelnorm, or other 5-HT4 agonists
  * Opiods/narcotic analgesics
  * Prokinetics
  * Serotonin re-uptake inhibitors or tricyclic antidepressants
  * Calcium antagonists
* Patients who are breastfeeding, pregnant, or intend to become pregnant during the study.
* Female patients of childbearing potential who refuse a pregnancy test.
* Patients with a known allergy to corn or polyethylene glycol.
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Patients who, within the past 30 days have participated in an investigational clinical study
* Patients that have undergone a colonoscopy within 30 days of beginning the 14 day observation period.
* Patients that are currently taking, or have previously been treated with polyethyleneglycol3350

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-08; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
A successful outcome is defined as no longer meeting the definition of constipation using ROME I criteria

SECONDARY OUTCOMES:
Analysis of individual ROME I criteria
Safety (adverse events and laboratory testing)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Herrera, MD, Principal Investigator — University of South Alabama
Locations (41):
- United States (41):
  - Hoover, Alabama
  - Mobile, Alabama
  - Pell City, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Sacramento, California
  - Washington D.C., District of Columbia
  - Kissimmee, Florida
  - Lake Worth, Florida
  - Largo, Florida
  - Ocoee, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Oakbrook Terrace, Illinois
  - Peoria, Illinois
  - Overland Park, Kansas
  - Laurel, Maryland
  - Springfield, Massachusetts
  - St Louis, Missouri
  - South Bound Brook, New Jersey
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Greer, South Carolina
  - Bristol, Tennessee
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia

REFERENCES:
- [Derived] Menees SB, Lembo AJ, Chey WD. Polyethylene Glycol 3350 in the Treatment of Chronic Idiopathic Constipation: Post hoc Analysis Using FDA Endpoints. Can J Gastroenterol Hepatol. 2022 Sep 9;2022:3533504. doi: 10.1155/2022/3533504. eCollection 2022. PMID 36120087